CLINICAL TRIAL: NCT06783894
Title: Elliptical Physical Activity and Sexual Dysfunction in Males With Irritable Bowel Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, Department of Physical Therapy for Cardiovascular/Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00014233-20
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Irritable Bowel Syndrome; Erectile Dysfunction
MeSH Terms: conditions — Irritable Bowel Syndrome; Erectile Dysfunction | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group I (Experimental): twenty irritable bowel syndrome men with sexual dysfunction ( weak erection of penis or erectile dysfunction) will perform ellpitical physical activity (40 minutes on elliptical trainer three times weekly. the duration of physical activity will be 12 weeks.
  Interventions: Behavioral: exercise (elliptical training)
- Group II (No Intervention): twenty irritable bowel syndrome men with sexual dysfunction (weak erection of penis or erectile dysfunction) will perform no type of activity (wait list group).

INTERVENTIONS:
Behavioral: exercise (elliptical training) — twenty irritable bowel syndrome men with sexual dysfunction ( weak erection of penis or erectile dysfunction) will perform ellpitical physical activity (40 minutes on elliptical trainer three times weekly. the duration of physical activity will be 12 weeks.
  Arms: group I

SUMMARY:
psychological disturbances resulting from irritable bowel syndrome causes sexual dysfunction in men such as weak erection of penis. The different exercise forms are important in improving symptoms of this syndrome and exercise also may improve sexual dysfunction in men

DETAILED DESCRIPTION:
Forty irritable bowel syndrome men with sexual dysfunction ( weak erection of penis or erectile dysfunction) will divided into Group I or Group II . The group will contain twenty subjects. Group I will perform ellpitical physical activity (40 minutes on elliptical trainer three times weekly. the duration of physical activity will be 12 weeks. Group II will not perform any physical activity.

ELIGIBILITY:
Inclusion Criteria:

* men with irritable bowel syndrome
* men with erectile dysfunction
* married men

Exclusion Criteria:

* obese men
* chest/renal disease men
* cardiac/metabolic disease men
* systemic disease men

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — based on self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2025-01-12 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-02 (Estimated)

PRIMARY OUTCOMES:
international index of erectile fucntion | it will be assessed after 12 weeks
  it is questionnaire that contains five questions assessing erectile functions

SECONDARY OUTCOMES:
Irritable Bowel Syndrome Severity Scoring System | it will be assessed after 12 weeks
  it is a questionnaire that assesses the severity symptoms related to irritable bowel syndrome
Irritable Bowel Syndrome Quality of Life Questionnaire | it will be assessed after 12 weeks
  it is a questionnaire that assesses the quality of life in patients irritable bowel syndrome
State Anxiety Inventory | it will be assessed after 12 weeks
  it is a questionnaire that assesses the long standing anxiety
Beck depression inventory | it will be assessed after 12 weeks
  it is a questionnaire that assesses depression symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ali MA Ismail, Principal Investigator — Cairo University
Locations (1):
- faculty of physical therapy Cairo university, Dokki, Giza Governorate, Egypt